CLINICAL TRIAL: NCT01780233
Title: A Single-dose Crossover Study of Fentanyl Sublingual Spray 400 Mcg Versus Actiq® 400 Mcg Versus Fentanyl Citrate Injection (iv) 100 Mcg Under Fasted Conditions
Brief Title: Pharmacokinetic Study of Fentanyl 400 µg Sublingual Spray, Actiq® 400 µg Transmucosally, and Fentanyl Citrate Injection 100 µg Intravenously (iv)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INS-06-003
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Fentanyl; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fentanyl 400 µg sublingual spray + naltrexone 50 mg (Experimental): Patients received a single administration of 400 µg of fentanyl spray sublingually + naltrexone hydrochloride 50 mg orally.
  Interventions: Drug: Fentanyl 400 µg sublingual spray; Drug: Naltrexone 50 mg
- Actiq® 400 µg transmucosally + naltrexone 50 mg (Active Comparator): Patients received a single administration of 400 µg of Actiq® transmucosally + naltrexone hydrochloride 50 mg orally.
  Interventions: Drug: Actiq® 400 µg transmucosally; Drug: Naltrexone 50 mg
- Fentanyl citrate injection 100 µg iv + naltrexone 50 mg (Active Comparator): Patients received a single administration of 100 µg of fentanyl citrate intravenously + naltrexone hydrochloride 50 mg orally.
  Interventions: Drug: Fentanyl citrate injection 100 µg intravenously; Drug: Naltrexone 50 mg

INTERVENTIONS:
Drug: Fentanyl 400 µg sublingual spray
  Arms: Fentanyl 400 µg sublingual spray + naltrexone 50 mg
Drug: Actiq® 400 µg transmucosally — Actiq® 400 µg is a solid formulation of fentanyl citrate on a plastic stick that dissolves slowly in the mouth for absorption across the buccal mucosa.
  Other Names: fentanyl citrate
  Arms: Actiq® 400 µg transmucosally + naltrexone 50 mg
Drug: Fentanyl citrate injection 100 µg intravenously
  Arms: Fentanyl citrate injection 100 µg iv + naltrexone 50 mg
Drug: Naltrexone 50 mg — Naltrexone hydrochloride was administered approximately 12 hours and 1 hour prior to and 12 hours after each dose of fentanyl to minimize the occurrence of unacceptable adverse effects (eg, decreased respiration, nausea) often associated with administration of fentanyl.

SUMMARY:
The objective of this study was to compare the rate of absorption and bioavailability of fentanyl 400 µg sublingual spray, Actiq® 400 µg transmucosally, and fentanyl citrate injection 100 µg intravenously.

DETAILED DESCRIPTION:
This was a Phase I, single-dose, open-label, randomized, 3-period, 3-treatment cross over study in which 21 healthy subjects received single doses of fentanyl 400 µg sublingual spray, Actiq® 400 µg transmucosally, and fentanyl citrate injection 100 µg intravenously following a 10-hour overnight fast. There was a 7 day washout period between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breast-feeding female between the ages of 18-55 inclusive.
* Body Mass Index (BMI) between 18-30 kg/m^2, inclusive, and body weight of at least 60 kg (132 lbs).
* Subject was healthy according to the medical history, laboratory results, and physical examination.

Exclusion Criteria:

* Had a presence or history of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition which, in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Had a clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at screening.
* Had a significant history of hypersensitivity to opioid analgesics, fentanyl or any related products, naltrexone, or severe hypersensitivity reactions (like angioedema) to any drugs.
* Had a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Had donated blood or plasma within 30 days prior to the first dose of study medication or during the course of this study.
* Had participated in another clinical trial within 30 days prior to the first dose of study medication or during the course of this study.
* Had used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication or during the course of this study.
* Had used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication or during the course of this study.
* Had used enzyme altering drugs such as barbiturates, corticosteroids, phenothiazines, cimetidine, carbamazepine, etc, within 30 days prior to the first dose of study medication or during the course of this study.
* Had used opioid analgesics within the last 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Time to reach the maximum drug concentration (Tmax) in plasma | Up to 60 minutes pre-dose to 36 hours post-dose

SECONDARY OUTCOMES:
Maximum drug concentration (Cmax) in plasma | Up to 60 minutes pre-dose to 36 hours post-dose
Area under the plasma concentration-time curve from time-0 to the time of the last quantifiable concentration (AUClast) | Up to 60 minutes pre-dose to 36 hours post-dose
Area under the plasma concentration-time curve from time-0 extrapolated to infinity (AUCinf) | Up to 60 minutes pre-dose to 36 hours post-dose
Percentage of AUCinf based on extrapolation (AUCextrap) | Up to 60 minutes pre-dose to 36 hours post-dose
Observed elimination rate constant (λz) | Up to 60 minutes pre-dose to 36 hours post-dose
Observed terminal elimination half-life (T1/2) | Up to 60 minutes pre-dose to 36 hours post-dose
Time of the last measurable concentration of drug (Tlast) in plasma | Up to 60 minutes pre-dose to 36 hours post-dose
Last quantifiable drug concentration (Clast) in plasma | Up to 60 minutes pre-dose to 36 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Neha Parikh, Study Director — INSYS Therapeutics Inc; Frederick A. Bieberdorf, MD, Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States

REFERENCES:
- [Derived] Parikh N, Goskonda V, Chavan A, Dillaha L. Single-dose pharmacokinetics of fentanyl sublingual spray and oral transmucosal fentanyl citrate in healthy volunteers: a randomized crossover study. Clin Ther. 2013 Mar;35(3):236-43. doi: 10.1016/j.clinthera.2013.02.017. PMID 23497761